CLINICAL TRIAL: NCT00497575
Title: Diagnosis and Follow-up of Patients With Subclinical Hypothyroidism
Acronym: CHRO1
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Other Study IDs: no. 2002C23037
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2007-07-06 (Estimated); Status verified 2007-07

CONDITIONS: Congenital Hypothyroidism; L-Thyroxine; Follow-Up
Keywords: Congenital Hypothyroidism; diagnosis; L-thyroxine; newborn screening
MeSH Terms: conditions — Congenital Hypothyroidism; Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Long term follow-up of the patients with delayed TSH elevation or subclinical hypothyroidism has been seldom reported. The purpose of this study was to explore the diagnostic criteria for subclinical hypothyroidism and the initial dosage of L-thyroxine through long-term follow up for infants with subclinical hypothyroidism ，and evaluate the curative effect.

DETAILED DESCRIPTION:
Long term follow-up of the patients with delayed TSH elevation or subclinical hypothyroidism has been seldom reported. The purpose of this study was to explore the diagnostic criteria for subclinical hypothyroidism and the initial dosage of L-thyroxine through long-term follow up for infants with hyperthyrotropinemia，and evaluate the curative effect.All live-born neonates in province took part in the screening program from October, 1999 to September ,2006. Laboratory tests are performed as a time resolved fluoro-immunoassay (TRFIA). TSH is measured with a cut-off > 9 mU/L. The diagnostic standard for subclinical hypothyroidism was: TSH ≥ 20 mU/L, T3 and T4 normal or low-normal ,or TSH > 5.6 mU/L and < 20 mU/L on initial determination and on follow-up or TSH levels increase on follow-up and/or gradually declining T4 levels.L-Thyroxine was administered for substitution therapy. After 2 years therapy，allround evaluation was performed. Compare the correlation to effects with different level of TSH、starting time of therapy and environment. Compare the effects between subclinical、temporary and permanent hypothyroidism.

ELIGIBILITY:
Inclusion Criteria:

* The diagnostic standard for manifest hypothyroidism and subclinical hypothyroidism was defined as follows:

  * Hypothyroidism - TSH > 40 mU/L and T3 and T4 below the reference range or TSH > 40 mU/L, T3 normal and T4 below the reference range [2]
  * Subclinical hypothyroidism - TSH ≥ 20 mU/L, T3 and T4 normal or low-normal or TSH > 5.6 mU/L and < 20 mU/L on initial determination and on follow-up or TSH levels increase on follow-up and/or gradually declining T4 levels.

Max Age: 5 Years | Sex: All
Age Groups: Child
Dates: Start 1999-10; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: zhengyan Zhao, doctor, Study Director — Pediatric Society of the Chinese Medical Association